CLINICAL TRIAL: NCT03685058
Title: The Effect of Light Curable Resin Modified Glass Ionomer Varnish on Inhibiting the Progression of Non-Cavitated Proximal Carious Lesions: A Randomized Controlled Trial
Brief Title: Effect of Light Curable Resin Modified Glass Ionomer Varnish on Non-Cavitated Proximal Carious Lesions' Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najlaa Alamoudi, Professor in Pediatric Dentistry Department, Medical Director, KAU-DH Program Director, Post Grad Studies for Master and PhD programs Program Director,of Saudi Commission for Health Specialities, Faculty of Dentistry- King Abdulaziz University, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAlamoudi
Record Dates: First submitted 2017-10-10; First posted 2018-09-26 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Dental Caries; Dental White Spot
Keywords: Initial caries treatment; Non-cavitated caries treatment; Incipient caries treatment; Proximal caries; Primary teeth; Light curable resin modified glass ionomer varnish; Vanish XT varnish; Clinpro XT varnish; Dental white spot lesions
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: The study design will be a split mouth, randomized controlled clinical trial in which the teeth will be randomly assigned to be either in the test group or control group in a 1:1 ratio.
  The control group: will be treated with standard-of-care preventive measures which includes application of 5% sodium fluoride (NaF) topical varnish, oral hygiene instruction, and dietary counseling.
  The test group: will be treated with light curable resin modified glass ionomer (RMGI) varnish in addition to standard-of-care preventive measures.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Because of the nature of the study, the investigator who will apply the treatment will not be blind to the group allocation of the lesion. Yet, the investigators who will evaluate the radiographs, DIAGNOcam images, and perform the visual examination will be blinded to which group the lesion they are evaluating belongs. In addition, the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- The control group (Active Comparator): A total of 88 non-cavitated proximal carious lesions treated with standard-of-care preventive measures which include application of 5% sodium fluoride topical varnish (Vanish 5% Sodium Fluoride White Varnish with Tri-Calcium Phosphate, 3M ESPE, St. Paul, MN, U.S.A.), oral hygiene instruction, and dietary counseling applied at initial, six-months follow-up, and 12-months follow-up visits.
  Interventions: Other: standard-of-care preventive measures
- The test group (Experimental): Intervention: A total of 88 non-cavitated proximal carious lesions treated with light curable resin modified glass ionomer varnish (Vanish™ XT Extended Contact Varnish, 3M ESPE, St. Paul, MN, U.S.A.) at initial and six-months follow-up visits. In addition to, standard-of-care preventive measures, applied at initial, six-months follow-up, and 12-months follow-up visits.
  Interventions: Device: Light curable resin modified glass ionomer varnish; Other: standard-of-care preventive measures

INTERVENTIONS:
Device: Light curable resin modified glass ionomer varnish — Treatment of non-cavitated proximal carious lesions with light curable resin modified glass ionomer varnish at initial and six-months follow-up visits, in addition, the patient will receive standard-of-care preventive measures, at initial, six-months follow-up, and 12-months follow-up visits.
  Other Names: Vanish™ XT Extended Contact Varnish
  Arms: The test group
Other: standard-of-care preventive measures — Patient will receive standard-of-care preventive measures which include application of 5% sodium fluoride topical varnish, oral hygiene instructions, and dietary counseling at initial, six-months follow-up, and 12-months follow-up visits

SUMMARY:
The standard-of-care preventive measures to stop early tooth decay from becoming worse is by fluoride application, diet counseling, and oral hygiene instructions. This standard way is not always successful. The purpose of this study is to compare standard-of-care preventive measures to stop further tooth decay to standard-of-care preventive measures in addition to a light curable resin modified glass ionomer (RMGI) varnish material (Vanish XT). The material is used for root surface sensitivity treatment, site specific protective coating for newly erupted teeth and other tooth surfaces including early tooth decay.

To be in this study the child must be five to eight years old, medically healthy, attending the Pediatric Dentistry Clinics in King Abdulaziz University Dental Hospital (KAUDH),diagnosed to have at least two primary molars and/ or first permanent molars with early-stage caries (using bitewing radiographs, near infrared digital imaging transilluminaton (NIDIT), and visual assessment), and willing to return for follow up visits. If the child is eligible and the parents agree to the participation of their child in this study, the researcher will review the child's personal and medical history.

The child's two included molars diagnosed with early-stage caries will be randomly assigned to one of two groups: Control Group: will receive standard-of-care preventive measures. Test Group: will receive RMGI varnish application plus the standard-of-care preventive measures. The child will be followed up at six months and 12 months. A dental examination will be done using the same methods used in the first examination to determine whether the caries has become deeper or not. The child may be withdrawn from the study at this point if the caries has become too deep and the tooth will then need a filling.

The child's medical status will be up-dated, reinforcement of oral hygiene instruction and diet counseling will be provided, and fluoride varnish application will be applied to all the teeth in both six and 12 months follow-ups.The RMGI varnish will be reapplied to the test teeth at the six months follow up.

DETAILED DESCRIPTION:
Materials and Methods Sample:It will be 88 contralateral matched primary molars and/or first permanent molars with non-cavitated proximal carious lesion to be treated in children attending the Pediatric Dentistry Clinics at KAUDH, Jeddah, Saudi Arabia.The included lesions will be randomly allocated in a split-mouth design to be either in the test group or control group:The control group: will be treated with standard-of-care preventive measures which includes application of 5% sodium fluoride (NaF) topical varnish (Vanish 5% Sodium Fluoride White Varnish with Tri-Calcium Phosphate, 3M ESPE, Dental product 44-0007-4718-6-B, St. Paul, MN, 55144-1000 U.S.A. ), oral hygiene instruction, and dietary counseling.The test group: will be treated with light curable RMGI varnish (Vanish™ XT Extended Contact Varnish, 3M ESPE, Dental product 44-0007-4718-6-B, St. Paul, MN, 55144-1000 U.S.A.) in addition to standard-of-care preventive measures.

The Sample size:It was calculated based on the assumptions of odds of caries prevention for the light curable RMGI varnish and the fluoride varnish will be 5.6 and 1.9 respectively based on the literature. The estimated sample is a minimum of 80 pairs (160 lesions) of non-cavitated proximal carious lesions in primary molars and/or first permanent molars are required by the end of the study to detect a statistical difference between the groups at significance level of 0.05 with a power of 80% the sample size was calculated using GPower 3.1 software .To compensate for loss to follow up or other causes of attrition, an additional 10% will be added to the sample size, thus eight pairs will be added with a total of 88 pairs (176 lesions) needed at the start of the study.

Materials and Equipment:

For the lesion diagnosis: Bitewing radiographic examination will be performed using an XCP extension cone paralleling system with photo-stimulable phosphor (PSP) plate biteblocks. The NIDIT examination will be performed using the DIAGNOcam device (DIAGNOcam 2170, Sn 1001941; Kavo). Clinical examination will be performed using mouth mirrors, Community Periodontal Index probe, dental floss without wax, orthodontic elastic separators, a plier for teeth separation for the visual examination, and dental chair light.

Consent and ethical approval:Approval will be obtained from King Abdulaziz University, Research Ethics Committee of the Faculty of Dentistry. The nature of the study will be explained to the parents of the children who meet the inclusion criteria. An informed written consent form will be obtained from all the parents who agree to have their children participate in the study.

Study design:The study design will be a split mouth,triple-blinded, randomized controlled clinical trial following CONSORT guidelines.The teeth will be randomly assigned to one of the two study groups in 1:1 ratio.

Recruitment of the Participants:

Children who are attending the Pediatric Dentistry Clinics in KAUDH during the years 2017 and 2018 over a period of three to six months, who fulfill the subject's inclusion criteria will be initially screened by the primary investigator using bitewing radiographs for the presence of at least two matched bilateral primary molars and/or first permanent molars with non-cavitated proximal carious lesion in the same surfaces. For children who meet all the inclusion criteria, a written consent will be obtained from their parents/guardians to allow their participation in the study. If the subject is diagnosed with more than one qualified pair of lesions, the pairs will be included in the study.

Personal and Medical Information:Before examination, the subject's medical history will be reviewed by the primary investigator along with the age, gender, and nationality.

Lesion Selection and Clinical Assessment:

Radiographic examination:The baseline screening bite-wing radiographs will be taken on both sides of the mouth of the participants . The radiographs will be assessed by two calibrated trained examiners using the following score system: 0: No radiolucency. E1: Radiolucency within outer half of the enamel. E2: Radiolucency in the inner half of the enamel. D1: Radiolucency in the outer third of the dentin. D2: Radiolucency in the middle third of the dentin. D3: Radiolucency in the inner third of the dentin. Disagreements between the first two examiners will be resolved by a third calibrated trained examiner.Teeth that are scored E1, E2, and D1 by two calibrated trained examiners will be included in the study.

Near Infrared Digital Imaging Transillumination: the tooth will be examined by two calibrated trained examiners using the DIAGNOcam according to manufacture instructions. The following scoring system will be used: 0: Sound surface.1: First visible sign of enamel caries. 2: Established enamel caries lesion.3: Established enamel caries lesion with an isolated spot reaching the EDJ.4: Dentin caries penetrating the EDJ lineary. 5: Deep dentin caries lesion. Disagreements between the first two examiners will be resolved by a third calibrated trained examiner. An orthodontic elastic separator will be placed in the corresponding interproximal area to facilitate the subsequent visual examination of the lesion after two days.

Visual Caries Assessment:The orthodontic elastic separators will be removed, and caries will be scored clinically by two calibrated trained examiners using the ICDAS II visual scoring system: 0:clinical sound surfaces 1 and 2: non-cavitated lesions (in 1 air-drying is required to see the lesion and in 2 the lesion is visible without air-drying). 3:Localized enamel breakdown due to caries with no visible dentin. 4:Underlying dark shadow from dentin with or without localized enamel breakdown. 5 and 6:increasing stages of dentine cavitation. Disagreements between the first two examiners will be resolved by a third calibrated trained examiner.Teeth that are scored one and two by two calibrated trained examiners will be included in the study.Other variables that will be recorded at this visit: (1) decayed, missing, filled permeant tooth due to caries (DMFT) and decayed, missing, filled primary tooth due to caries (dmft) score ; (2) plaque score of the included teeth at the time of teeth treatment ; (6) presence of gingival bleeding at the included interproximal site at the time of tooth treatment; (7) and the restoration status of adjacent surface.

Treatment of Lesions: The test group: the lesions will be treated with Vanish XT varnish according to the manufacturer's instructions.

The control group: the lesion will be treated with the Vanish 5% NaF White Varnish according to the manufacturer's instructions. To blind the patient and the parents to which treatment is done to the control tooth, a simulation of the light curable RMGI varnish application will be done, i.e. a thin layer of the fluoride varnish will be applied to the control tooth surface and the light-cure will be held for 20 seconds without turning it on for the purpose of blinding. Then all the teeth will receive an application of the 5% NaF varnish as part of standard of care preventive measures along with oral hygiene instruction and diet counseling.

Follow-up The included subjects will be followed up at six and 12 months for clinical, radiographic, and NIDIT evaluation. At the six months' follow up, the light curable RMGI varnish will be applied in the test group lesions. All the teeth in both groups (test and control) will receive 5% NaF varnish application, along with reinforcement of oral hygiene instruction and diet counseling will be provided.every 6 months. At the six and 12 months follow ups, the subjects will be re-examined as at baseline by two calibrated trained examiners who will be blinded to which treatment group the lesion belongs. Disagreements between the first two examiners will be resolved by a third calibrated blinded examiner. If two of the examiners agree that there is no caries progression, the lesion will be regarded as an arrested lesion. If they agree that there is caries progression, the lesion will be regarded as to have progressed.

Randomization:The subjects will be included after at least one pair of qualified non-cavitated proximal carious lesion meeting the inclusion criteria are identified. Then randomization for the materials for both sides will be done.To ensure the balance of the treatment materials in both sides, block randomization will be generated, different sequence will be randomized for subjects according to the number of molar pairs that will be included in the study in that subject.

Training in the Caries Recording Systems:Inter-examiner and intra-examiner calibration will be done for radiographic, clinical and DIAGNOcam by calibrated examiners. Intra-examiner calibration will be done for DMFT/dmft index. Training will be done until the desired inter- and intra-examiner agreement is achieved.

Statistical analysis:The data will be collected and statistically analyzed using Windows IBM SPSS (Version 22). A P value of < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

The subject's inclusion criteria:

The child has at least two matched bilateral primary molars and/or first permanent molars with proximal carious lesions in the same surfaces in enamel or outer dentin third as by bitewing radiographic examination and are non-cavitated by visual examination.

* Their ages are five to eight years.
* Healthy.
* No known allergies to any of the components of the dental materials used in the study.
* The parents are willing to commit to the follow-up visits.
* Child is generally cooperative for dental treatment.

The tooth's inclusion criteria:

1. Primary molar and/or first permanent molars with a proximal carious lesion in enamel or outer dentin third assessed by bitewing radiographic examination and that is found to be non-cavitated after ICDAS visual examination.
2. Presence of a tooth adjacent to the lesion.
3. Normal tooth structure.
4. Absence of tooth mobility.
5. Tooth does not require restorative treatment.

Exclusion Criteria:

•The subject's exclusion criteria:

* Children with a medical history of a chronic disease.
* Children who have abnormalities that affect tooth structure.
* The need of sedation or general anesthesia for dental treatment.

The tooth exclusion criteria:

* Primary molar and/or first permanent molars with a proximal carious lesion extending beyond the outer dentin third assessed by bitewing radiographic examination.
* Primary molar and/or first permanent molars with a proximal carious lesion that is cavitated assessed by ICDAS visual examination.
* Non-cavitated proximal carious lesion on the mesial of the first primary molars because the contact area with the primary canine is narrow and the possible presence of the primate space.
* Distal surfaces of the first permanent molars because there is no contact with the second permanent molar (does not erupt in this age group).

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Clinical progression of non-cavitated proximal carious lesions measured using ICDAS six months after treatment | After six of treatment
  To evaluate the clinical progression of non-cavitated proximal carious lesions in primary molars and first permanent molars measured using the ICDAS after treatment with light curable RMGI varnish in addition to standard-of-care preventive measures compared to standard-of-care preventive measures alone after six months.
Clinical progression of non-cavitated proximal carious lesions measured using ICDAS 12 months after treatment | After 12 months.
  To evaluate the clinical progression of non-cavitated proximal carious lesions in primary molars and first permanent molars measured using the ICDAS after treatment with light curable RMGI varnish in addition to standard-of-care preventive measures compared to standard-of-care preventive measures alone after 12 months.
Radiographic progression of non-cavitated proximal carious lesions assessed using bitewing radiographs six months after treatment | After six months
  To evaluate the radiographic progression of non-cavitated proximal carious lesions in primary molars and first permanent molars assessed by examination of bitewing radiographs after treatment with light curable RMGI varnish in addition to standard-of-care preventive measures compared to standard-of-care preventive measures alone after six months.
Radiographic progression of non-cavitated proximal carious lesions assessed using bitewing radiographs 12 months after treatment | After 12 months
  To evaluate the radiographic progression of non-cavitated proximal carious lesions in primary molars and first permanent molars assessed by examination of bitewing radiographs after treatment with light curable RMGI varnish in addition to standard-of-care preventive measures compared to standard-of-care preventive measures alone after 12 months.
Progression of non-cavitated proximal carious lesions measured with NILT six months after treatment | After six months
  To evaluate the progression of non-cavitated proximal carious lesions in primary molars and first permanent molars measured with NILT after treatment with light curable RMGI varnish in addition to standard-of-care preventive measures compared to standard-of-care preventive measures alone after six months.
Progression of non-cavitated proximal carious lesions measured with NILT 12 months after treatment | After 12 months
  To evaluate the progression of non-cavitated proximal carious lesions in primary molars and first permanent molars measured with NILT after treatment with light curable RMGI varnish in addition to standard-of-care preventive measures compared to standard-of-care preventive measures alone after 12 months.

SECONDARY OUTCOMES:
The effect of plaque accumulation on the success rate of the treatment | After 12 months
  To evaluate the effect of plaque accumulation on the success rate of light curable RMGI varnish and standard-of-care preventive measures in inhibiting the progression of non-cavitated proximal carious lesions in comparison to standard of care preventive measures only.
The effect of gingival inflammation on the success rate of the treatment | After 12 months
  To evaluate the effect of gingival inflammation on the success rate of light curable RMGI varnish and standard-of-care preventive measures in inhibiting the progression of non-cavitated proximal carious lesions in comparison to standard of care preventive measures only.
he effect of the presence of adjacent restoration on the success rate of the treatment | After 12 months
  To evaluate the effect of the presence of adjacent restoration on the success rate of light curable RMGI varnish and standard-of-care preventive measures in inhibiting the progression of non-cavitated proximal carious lesions in comparison to standard of care preventive measures only.
The effect of caries severity on the success rate of the treatment | After 12 months
  To evaluate the effect of caries severity on the success rate of light curable RMGI varnish and standard-of-care preventive measures in inhibiting the progression of non-cavitated proximal carious lesions in comparison to standard of care preventive measures only.

CONTACTS AND LOCATIONS:
Overall Officials: Najlaa M Alamoudi, BDS,MSc,DSc, Principal Investigator — King Abdulaziz University, Faculty of Dentistry
Locations (1):
- King abulaziz University, Dental University Hospital, Jeddah, P.O Box 80209, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehta A, Paramshivam G, Chugh VK, Singh S, Halkai S, Kumar S. Effect of light-curable fluoride varnish on enamel demineralization adjacent to orthodontic brackets: an in-vivo study. Am J Orthod Dentofacial Orthop. 2015 Nov;148(5):814-20. doi: 10.1016/j.ajodo.2015.05.022. PMID 26522042
- [Background] Young DA, Novy BB, Zeller GG, Hale R, Hart TC, Truelove EL; American Dental Association Council on Scientific Affairs; American Dental Association Council on Scientific Affairs. The American Dental Association Caries Classification System for clinical practice: a report of the American Dental Association Council on Scientific Affairs. J Am Dent Assoc. 2015 Feb;146(2):79-86. doi: 10.1016/j.adaj.2014.11.018. PMID 25637205
- [Background] Anusavice KJ. Present and future approaches for the control of caries. J Dent Educ. 2005 May;69(5):538-54. PMID 15897335
- [Background] Sochtig F, Hickel R, Kuhnisch J. Caries detection and diagnostics with near-infrared light transillumination: clinical experiences. Quintessence Int. 2014 Jun;45(6):531-8. doi: 10.3290/j.qi.a31533. PMID 24618570
- [Background] Ekstrand KR, Martignon S, Ricketts DJ, Qvist V. Detection and activity assessment of primary coronal caries lesions: a methodologic study. Oper Dent. 2007 May-Jun;32(3):225-35. doi: 10.2341/06-63. PMID 17555173
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Background] Weyant RJ, Tracy SL, Anselmo TT, Beltran-Aguilar ED, Donly KJ, Frese WA, Hujoel PP, Iafolla T, Kohn W, Kumar J, Levy SM, Tinanoff N, Wright JT, Zero D, Aravamudhan K, Frantsve-Hawley J, Meyer DM; American Dental Association Council on Scientific Affairs Expert Panel on Topical Fluoride Caries Preventive Agents. Topical fluoride for caries prevention: executive summary of the updated clinical recommendations and supporting systematic review. J Am Dent Assoc. 2013 Nov;144(11):1279-91. doi: 10.14219/jada.archive.2013.0057. PMID 24177407
- [Background] Guideline on Caries-risk Assessment and Management for Infants, Children, and Adolescents. Pediatr Dent. 2016 Oct;38(6):142-149. No abstract available. PMID 27931452
- [Background] Espelid I, Tveit AB. Clinical and radiographic assessment of approximal carious lesions. Acta Odontol Scand. 1986 Feb;44(1):31-7. doi: 10.3109/00016358609041295. PMID 3456691
- [Background] Martignon S, Ekstrand KR, Ellwood R. Efficacy of sealing proximal early active lesions: an 18-month clinical study evaluated by conventional and subtraction radiography. Caries Res. 2006;40(5):382-8. doi: 10.1159/000094282. PMID 16946605
- [Background] Bagher SM, Hegazi FM, Finkelman M, Ramesh A, Gowharji N, Swee G, Felemban O, Loo CY. Radiographic Effectiveness of Resin Infiltration in Arresting Incipient Proximal Enamel Lesions in Primary Molars. Pediatr Dent. 2018 May 15;40(3):195-200. PMID 29793566
- [Derived] Felemban OM, Khan JA, Alamoudi NM, El-Ashiry EA, Bagher SM. Perception of Pain With Bitewing, DIAGNOcam, and Teeth Separation Amongst Children. Int Dent J. 2024 Jun;74(3):631-637. doi: 10.1016/j.identj.2023.11.002. Epub 2024 Jan 12. PMID 38216389